CLINICAL TRIAL: NCT02403063
Title: Electromyographic Activity of the Diaphragm and of the Rectus Abdominis and Intercostal Muscles During Neostigmine, Sugammadex, or Neostigmine-sugammadex Enhanced Recovery After Neuromuscular Blockade With Rocuronium. A Randomised Controlled Study in Healthy Volunteers
Brief Title: Electromyographic Activity of the Respiratory Muscles During Neostigmine or Sugammadex Enhanced Recovery After Neuromuscular Blockade
Acronym: REDNESII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Guy CAMMU, MD, PhD, Anesthesiologist, Onze Lieve Vrouw Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TSGC03
Record Dates: First submitted 2015-03-17; First posted 2015-03-31 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Respiratory Muscles; Electromyography
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sugammadex (Active Comparator): Selective relaxant binding agent
  Interventions: Drug: Sugammadex
- neostigmine (Active Comparator): Acetylcholinesterase inhibitor
  Interventions: Drug: Neostigmine
- neostigmine-sugammadex (Experimental): Acetylcholinesterase inhibitor followed by a selective relaxant binding agent
  Interventions: Drug: Neostigmine-sugammadex

INTERVENTIONS:
Drug: Sugammadex — Administration of sugammadex 2mg/kg for enhanced recovery after neuromuscular blockade with rocuronium
  Other Names: Bridion
  Arms: sugammadex
Drug: Neostigmine — Administration of neostigmine 50µg/kg for enhanced recovery after neuromuscular blockade with rocuronium
  Other Names: Robinul-neostigmine
  Arms: neostigmine
Drug: Neostigmine-sugammadex — Administration of neostigmine 50µg/kg followed 3 minutes later by administration of sugammadex 2mg/kg for enhanced recovery after neuromuscular blockade with rocuronium
  Arms: neostigmine-sugammadex

SUMMARY:
It was recently shown that neostigmine reversal was associated with increased atelectasis and that high-dose neostigmine was associated with longer postoperative length of stay and with an increased incidence of pulmonary edema and reintubation. These study results were consistent with findings from a previous epidemiological study which revealed an absence of beneficial effects of neostigmine on postoperative oxygenation and reintubation. In our previous study, the effects of neostigmine / glycopyrrolate and sugammadex on the electromyographic activity of the diaphragm showed beneficial effects for sugammadex. This could be explained by a possible effect on neuromuscular transmission at the muscle level, but can also be explained by a neostigmine-induced decrease in total nerve activity. In a study in cats, neostigmine has been shown to reduce efferent phrenic nerve activity. The investigators aim to show a difference in phrenic nerve activity between neostigmine and sugammadex, administered alone or in combination, in healthy male volunteers.

DETAILED DESCRIPTION:
An auxiliary surface EMG will be recorded via ordinary skin electrodes at the diaphragm, and intercostal and rectus abdominis muscles. The degree of neuromuscular blockade is continuously measured by accelerometry of the adductor pollicis muscle with ulnar nerve stimulation (TOF-watch SX®). Anesthesia is induced with propofol and remifentanil. Manually assisted ventilation with an air/oxygen mixture of 40% oxygen is started as soon as patients are becoming apnoeic. Train-of-four (TOF) monitoring starts after the induction of anesthesia (before rocuronium administration) and continues until awakening. The investigators will insert a 16 Fr. nasogastric catheter which allows electrical activity of the diaphragm (Edi) registration (NAVA, Maquet, Solna, Sweden). After baseline measurements, 0.6 mg/kg rocuronium is injected. After tracheal intubation, subjects will be ventilated by a standard ventilation mode (tidal volume 7 ml/kg, frequency of 12 breaths per minute, inspired oxygen fraction of 30%), with end-tidal PCO2 targets of 30-35 mmHg and a PEEP of 5 cmH2O. SpO2 values will be maintained at ≥98%. Spontaneous recovery is allowed to progress until the re-appearance of the second twitch of the TOF. The volunteers will then receive either sugammadex 2mg/kg or neostigmine 50µg/kg + glycopyrrolate 10µg/kg (using the commercially available 5:1 co-formulation) or neostigmine 50µg/kg followed 3 minutes later by administration of sugammadex 2mg/kg. At the onset of spontaneous respiration, an arterial blood gas sample will be drawn. NAVA catheter positioning will be confirmed using the 'Edi catheter positioning' tool as soon as a signal is received. A second arterial blood gas sample will be drawn at the moment of awakening.

Diaphragm electromyographic activity (Edi, obtained from the NAVA catheter), airway pressure and flow are acquired at 100 Hz from the ventilator via an interface connected to a computer using commercially available software (Maquet Critical Care, Solna, Sweden). The auxiliary surface EMG will be recorded with a dedicated device (Dipha16, InBiolab, Groningen, The Netherlands) at the diaphragm, and intercostal and rectus abdominis muscles. All data will be stored and later analysed.

ELIGIBILITY:
Inclusion Criteria:

* Only male, healthy volunteers will be enrolled after an in-depth interview.
* Each participant must have the mental capacity to decide whether he takes part in the trial or not. Each participant must voluntarily give his written informed consent.
* Each participant must be between 18 and 40 years of age.
* Each participant must meet the American Society of Anaesthesiologists class I criteria.

Exclusion Criteria:

* The participant is known or suspected to have a neuromuscular disorder.
* The participant is known or suspected to have an allergic reaction to sugammadex, rocuronium, anaesthetic medications, or any drugs used during general anaesthesia.
* The participant is known or suspected to have an anatomical malformation impeding a proper intubation.
* The participant is known or suspected to have a history of malignant hyperthermia.
* The participant is known to have a renal insufficiency .
* The participant is known or suspected to have a chronic obstructive pulmonary disease GOLD classification 2 or higher.
* The participant is known to have an infection of the upper or lower airways, as diagnosed by clinical findings.

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Electromyographic activity of the respiratory muscles during recovery enhanced by sugammadex, neostigmine or neostigmine followed by sugammadex | Participants will be followed from administration of study drug until tracheal extubation, an expected average of 1 hour
  EMG activity of the diaphragm (EMGdi), and of the rectus abdominis and of the intercostal muscles during recovery enhanced by sugammadex 2mg/kg or neostigmine 50µg/kg or neostigmine 50µg/kg followed 3 minutes later by administration of sugammadex 2mg/kg

SECONDARY OUTCOMES:
Tidal volume of breaths recorded by the ventilator | Participants will be followed from administration of study drug until tracheal extubation, an expected average of 1 hour
The partial pressure of O2 and of carbon dioxide in arterial blood | Participants will be followed from administration of study drug until tracheal extubation, an expected average of 1 hour
The arterial oxygen saturation | Participants will be followed from induction of anesthesia until two hours after extubation of the trachea, an expected average of 3 hours
  Saturation of hemoglobin with oxygen as measured by Pulse Oximetry

CONTACTS AND LOCATIONS:
Overall Officials: GUY CAMMU, MD, PhD, Principal Investigator — OLV Hospital, Aalst, Belgium
Locations (1):
- OLV Hospital, Aalst, Belgium

REFERENCES:
- [Background] Sasaki N, Meyer MJ, Malviya SA, Stanislaus AB, MacDonald T, Doran ME, Igumenshcheva A, Hoang AH, Eikermann M. Effects of neostigmine reversal of nondepolarizing neuromuscular blocking agents on postoperative respiratory outcomes: a prospective study. Anesthesiology. 2014 Nov;121(5):959-68. doi: 10.1097/ALN.0000000000000440. PMID 25225821
- [Background] Eikermann M, Fassbender P, Malhotra A, Takahashi M, Kubo S, Jordan AS, Gautam S, White DP, Chamberlin NL. Unwarranted administration of acetylcholinesterase inhibitors can impair genioglossus and diaphragm muscle function. Anesthesiology. 2007 Oct;107(4):621-9. doi: 10.1097/01.anes.0000281928.88997.95. PMID 17893459
- [Background] Herbstreit F, Zigrahn D, Ochterbeck C, Peters J, Eikermann M. Neostigmine/glycopyrrolate administered after recovery from neuromuscular block increases upper airway collapsibility by decreasing genioglossus muscle activity in response to negative pharyngeal pressure. Anesthesiology. 2010 Dec;113(6):1280-8. doi: 10.1097/ALN.0b013e3181f70f3d. PMID 20980910
- [Background] Meyer MJ, Bateman BT, Kurth T, Eikermann M. Neostigmine reversal doesn't improve postoperative respiratory safety. BMJ. 2013 Mar 19;346:f1460. doi: 10.1136/bmj.f1460. No abstract available. PMID 23512446
- [Background] Schepens T, Cammu G, Saldien V, De Neve N, Jorens PG, Foubert L, Vercauteren M. Electromyographic activity of the diaphragm during neostigmine or sugammadex-enhanced recovery after neuromuscular blockade with rocuronium: a randomised controlled study in healthy volunteers. Eur J Anaesthesiol. 2015 Jan;32(1):49-57. doi: 10.1097/EJA.0000000000000140. PMID 25111539
- [Background] Fleming NW, Henderson TR, Dretchen KL. Mechanisms of respiratory failure produced by neostigmine and diisopropyl fluorophosphate. Eur J Pharmacol. 1991 Mar 19;195(1):85-91. doi: 10.1016/0014-2999(91)90384-3. PMID 2065714
- [Derived] Cammu G, Schepens T, De Neve N, Wildemeersch D, Foubert L, Jorens PG. Diaphragmatic and intercostal electromyographic activity during neostigmine, sugammadex and neostigmine-sugammadex-enhanced recovery after neuromuscular blockade: A randomised controlled volunteer study. Eur J Anaesthesiol. 2017 Jan;34(1):8-15. doi: 10.1097/EJA.0000000000000543. PMID 27902641